CLINICAL TRIAL: NCT06657248
Title: Prospective, Multicenter Study Evaluating the Midterm Clinical Performance and Safety of the Unicompartmental Univation® XF Pro Knee Implant
Brief Title: Clinical Performance and Safety of the Unicompartmental Univation® XF Pro Implant
Acronym: UNI_XF_PRO
Status: Not yet recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-22003
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gonarthritis; Degenerative Disease
Keywords: Degenerative medial unicompartmental Gonarthrosis; Unicompartmental knee arthroplasty; Safety and Performance
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- univation® XF Pro: Primary medial unicompartmental knee arthroplasty treated with implantation of unicompartmental knee prosthesis univation® XF Pro
  Interventions: Device: univation® XF Pro

INTERVENTIONS:
Device: univation® XF Pro — Primary medial unicompartmental knee arthroplasty
  Other Names: Unicompartmental knee arthroplasty

SUMMARY:
The study is designed as a prospective, observational, mid-term, multi-center follow-up study. It is planned to include 150 patients from 4 different study centres in Germany.

DETAILED DESCRIPTION:
The product under investigation is used in routine clinical practice and according to the authorized Instructions for Use (IfU). The data that is obtained in routine clinical use will be documented in an electronical Case Report Form (eCRF). The study's main purpose is the collection of clinical data on the safety and performance of the redesigned univation® XF Pro implant.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a primary medial unicompartmental knee endoprosthesis

Acc. to Instructions for Use:

* Both cruciate ligaments intact
* Lateral ligaments intact
* Leg axis amenable to passive correction
* Varus deformity under 15°
* Bending capability of at least 90°
* Extension deficit no greater than 5-10°
* Written informed consent of patient
* Kellgran & Lawrence Score > II (only straight or varus
* Patients with moderate radiological symptoms
* Patients without clinical symptoms

Exclusion Criteria:

* Pregnancy
* Patient age <18 and > 75 years
* BMI ≥ 40
* High risk patients ASA > III

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 75 years of age with an indication for a primary medial unicompartmental knee endoprosthesis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Functional patient-reported outcome | 5 years post-op
  The Oxford Knee Score (OKS) is a reliable 12-item, patient-reported questionnaire originally developed and validated specifically to assess function and pain in patients undergoing total knee replacement. It is short, reproducible, valid and sensitive to clinically important changes over time. Each of the 12 questions on the OKS is scored in the same way with the score decreasing as the reported symptoms increase (i.e. become worse). All questions are laid out with response categories denoting least (or no) symptoms to the left of the page (scoring 4) and those representing greatest severity lying on the right hand side (scoring 0), as detailed for question 1 below. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome.

SECONDARY OUTCOMES:
Implant survival [Kaplan-Meier] | until 5 years postoperatively
  Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period.
Quality of Life [EQ-5D-5L] compared to baseline | Preoperatively (baseline) and 3 months, 1 year, 2 years, 5 years postoperatively
  The 5-dimension 5-level measure of the health status, developed by the EuroQol Group (EQ-5D-5L) is a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
  The answer of each of the five dimensions result in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Progress of Clinical Outcome [Forgotten Joint Score-12] over follow-up period | 3 months, 1 year, 2 years, 5 years postoperatively
  The Forgotten Joint Score-12 (FJS-12) Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. These Patient Reported Outcome (PRO) questionnaires focus on patients' awareness of a specific joint in everyday life. In 12 Items the awareness for the artificial joint is assessed by the patient, each on a five point scale (Never / Almost Never / Seldom / Sometimes / Mostly) The Forgotten Joint Score assessment consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Radiological assessment: axis alignment (long leg x-ray) over time | at discharge (approx. 7-10 days postoperatively), 3 months, 1 year, 2 years, 5 years postoperatively
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. The radiographic evaluation of Alignment is based on long-leg x-rays
Radiological assessment: comparison of tibial slope over time | at discharge (approx. 7-10 days postoperatively), 3 months, 1 year, 2 years, 5 years postoperatively
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. Any changes of Tibial slope over the follow-up period is documented in the radiographic evaluation
Radiological assessment: Patella x-ray | at discharge (approx. 7-10 days postoperatively), 3 months, 1 year, 2 years, 5 years postoperatively
Number of Adverse events / serious adverse events over time | During the course of the study up to 5 years postoperatively
  During the course of the study, any upcoming intra- or postoperative (serious) adverse events (AE / SAE) or device effects related or not related to the product under investigation or the procedure, will be documented in the dedicated Case Report Forms. The total number of AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product
Number of Participants with radiological complications over time | During the course of the study up to 5 years postoperatively
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. All radiologically evident complications (including fracture, wear, loosening or radiolucencies) are cumulatively documented over the period of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Haaker, Prof. Dr., Principal Investigator — St. Vincenz Hospital Brakel
Locations (4):
- Germany (4):
  - Oberlinklinik gGmbH, Potsdam, Brandenburg
  - Lukas Krankenhaus, Bünde, North Rhine-Westphalia
  - St. Vincenz Hospital Brakel, Brakel
  - LMU Großhadern, München